CLINICAL TRIAL: NCT05308290
Title: Optimizing Cerebral Autoregulation During Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00137091; K76AG057020 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hip Fractures; Hip Arthropathy; Surgery; Delirium
MeSH Terms: conditions — Hip Fractures; Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood pressure managed by cerebral autoregulation (Experimental): In this arm cerebral autoregulation monitoring will be used to determine the lower and upper limits of cerebral autoregulation. Monitoring will continue throughout the surgery. Blood pressure management will be maintained to be within the limits of cerebral autoregulation.
  Interventions: Other: Blood pressure management according to cerebral autoregulation
- Standard of care blood pressure management (Active Comparator): In this arm cerebral autoregulation monitoring will be used for observation. The anesthesia provider will use usual care guidelines for blood pressure management.
  Interventions: Other: Blood pressure management according to usual care

INTERVENTIONS:
Other: Blood pressure management according to cerebral autoregulation — Intraoperative blood pressure will be targeted based on limits of cerebral autoregulation.
  Arms: Blood pressure managed by cerebral autoregulation
Other: Blood pressure management according to usual care — Intraoperative blood pressure will be targeted based on usual care.
  Arms: Standard of care blood pressure management

SUMMARY:
The purpose of this study is to conduct a pilot trial to determine the feasibility, safety, and potential efficacy of targeting mean arterial blood pressure (MAP) within the limits of cerebral autoregulation during surgery compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* planned hip or knee surgery (either for fracture or elective) or lung surgery
* age ≥60
* ambulatory at baseline
* expected duration of surgery > 90 minutes

Exclusion Criteria:

* Planned concurrent surgery
* Allergy to adhesive tape
* Short Blessed Test score >20
* Clinical diagnosis of dementia
* Opinion of either the anesthesiologist or surgeon that the patient is not appropriate.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Brown, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 patients were excluded during secondary screen before randomization
Period: Overall Study
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Started | 18 | 7
Completed | 15 | 5
Not Completed | 3 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — still in study followup | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 patients were excluded prior to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management | Total
Number analyzed (Participants) | 18 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.2) | 71.6 (7.8) | 70.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 7 | 25
Chronic Obstructive Pulmonary Disorder (COPD) [Count of Participants; unit: Participants] | 1 | 3 | 4
Diabetes Mellitus [Count of Participants; unit: Participants] | 4 | 3 | 7
Coronary Artery Disease [Count of Participants; unit: Participants] | 3 | 2 | 5
Cardiac Arrhythmia [Count of Participants; unit: Participants] | 1 | 1 | 2
Past Stroke or Transient Ischemic Attack [Count of Participants; unit: Participants] | 1 | 0 | 1
Hypertension [Count of Participants; unit: Participants] | 14 | 5 | 19
Hemoglobin (g/dl) [Mean (Standard Deviation); unit: (g/dl)] | 13.2 (1.6) | 13.7 (0.7) | 13.3 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure Outside Limits of Cerebral Autoregulation
Description: Extent (mmHg * hours) of mean arterial pressure outside limits of cerebral autoregulation after establishment of target mean arterial pressure.
Time Frame: Intraoperative, up to 5 hours
Population: Signals did not work with one participant and no data was collected.
Measure: Mean (Standard Deviation); unit: mmHg * hours
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Number analyzed (Participants) | 17 | 7
mmHg * hours | 2.2 (2.1) | 1.8 (1.2)
Statistical Analysis 1: Comparison: Blood Pressure Managed by Cerebral Autoregulation vs Standard of Care Blood Pressure Management; Test type: Other; p = 0.60, t-test, 2 sided — the a priori threshold for statistical significance was <0.05

2. Primary Outcome: Estimated Blood Loss
Description: Blood loss during surgery (mL).
Time Frame: Intraoperative, up to 5 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Number analyzed (Participants) | 18 | 7
mL | 17.5 (17.8) | 12.9 (19.8)
Statistical Analysis 1: Comparison: Blood Pressure Managed by Cerebral Autoregulation vs Standard of Care Blood Pressure Management; Test type: Other; p = 0.60, t-test, 2 sided — the a priori threshold for statistical significance was <0.05

3. Primary Outcome: Number of Participants With New Myocardial Infarction After Surgery
Description: Clinically diagnosed new myocardial infarction after surgery as a measure of incidence.
Time Frame: In the hospital after surgery, up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Number analyzed (Participants) | 18 | 7
Participants | 0 | 0
Statistical Analysis 1: Comparison: Blood Pressure Managed by Cerebral Autoregulation vs Standard of Care Blood Pressure Management; Test type: Other; p = 1.0, Fisher Exact — the a priori threshold for statistical significance was <0.05

4. Primary Outcome: Number of Participants With New Stroke After Surgery
Description: Clinically diagnosed new stroke after surgery as a measure of incidence.
Time Frame: In the hospital after surgery, up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Number analyzed (Participants) | 18 | 7
Participants | 0 | 0
Statistical Analysis 1: Comparison: Blood Pressure Managed by Cerebral Autoregulation vs Standard of Care Blood Pressure Management; Test type: Other; p = 1.0, Fisher Exact — the a priori threshold for statistical significance was <0.05

5. Secondary Outcome: Number of Participants That Develop Delirium After Surgery
Description: Development of delirium after surgery as diagnosed by the 3-Minute, Diagnostic Interview for Confusion Assessment Method (3D-CAM) or CAM-ICU.
Time Frame: In the hospital during the first 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
Number analyzed (Participants) | 18 | 7
Participants | 0 | 1
Statistical Analysis 1: Comparison: Blood Pressure Managed by Cerebral Autoregulation vs Standard of Care Blood Pressure Management; Test type: Other; p = 0.28, Fisher Exact — the a priori threshold for statistical significance was <0.05

6. Secondary Outcome: Change in General Cognitive Function as Assessed by the Short Blessed Test
Description: Will be assessed via Short Blessed Test. Scores range from 0-28 with 0 indicating no cognitive impairment and 28 indicating severe cognitive impairment.
Time Frame: Approximately 60, 180, and 365 Days after Surgery
Reporting Status: Not Posted

7. Secondary Outcome: Change in Executive Cognitive Function as Assessed by the Oral Trail Making Test
Description: Will be assessed via Oral Trail Making Test. The test is timed, and shorter times indicate better performance and longer times indicate worse performance.
Time Frame: Approximately 60, 180, and 365 Days after Surgery
Reporting Status: Not Posted

8. Secondary Outcome: Dementia Screening as Assessed by the AD8 Test
Description: Will be assessed via the Eight-item Interview to Differentiate Aging and Dementia Test (AD8). Scores range from 0-8 with 0 indicating no cognitive impairment and 8 indicating severe cognitive impairment consistent with dementia
Time Frame: 365 Days after Surgery
Reporting Status: Not Posted, anticipated posting 2026-07

9. Secondary Outcome: Change in General Overall Health and Disability as Assessed by the WHO Disability Assessment Schedule 2.0
Description: Will be assessed via the World Health Organization (WHO) Disability Assessment Schedule 2.0 (WHO-DAS 2.0). Scores range from 0-100 with 0 indicating no disability and 100 indicating severe disability.
Time Frame: Approximately 60, 180, and 365 Days after Surgery
Reporting Status: Not Posted

10. Secondary Outcome: Change in General Function as Assessed by the Instrumental Activities of Daily Living Questionnaire
Description: Score on Instrumental Activities of Daily Living. Scores range from 0-8, with 0 indicating severe impairment and 8 indicating no impairment.
Time Frame: Approximately 60, 180, and 365 Days after Surgery
Reporting Status: Not Posted

11. Secondary Outcome: Change in Ability to Ambulate Without Human Assistance
Description: Inability to walk more than 10 feet without human assistance.
Time Frame: Approximately 60, 180, and 365 Days after Surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 13-months
Arm/Group | Blood Pressure Managed by Cerebral Autoregulation | Standard of Care Blood Pressure Management
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 8/18 | 3/7
Other Adverse Events (participants affected / at risk) | 6/18 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blood Pressure Managed by Cerebral Autoregulation (N=18) | Standard of Care Blood Pressure Management (N=7)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hematuria or UTI (Renal and urinary disorders) | 1 (2) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blood Pressure Managed by Cerebral Autoregulation (N=18) | Standard of Care Blood Pressure Management (N=7)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pneumothorax prolonged (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subcutaneous Emphysema (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Delirium (Nervous system disorders) | 1 (1) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05308290/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT05308290/ICF_001.pdf